CLINICAL TRIAL: NCT03309787
Title: A Pilot Study of an eHealth-delivered Health Coaching Intervention
Brief Title: Health Coaching & Technology in a Weight Loss Center
Status: Completed | Type: Observational
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, John A. Batsis, MD, Associate Professor of Medicine and The Dartmouth Institute for Health Policy & Clinical Practice, Dartmouth-Hitchcock Medical Center
Other Study IDs: D17123
Record Dates: First submitted 2017-10-06; First posted 2017-10-16 (Actual); Results first posted 2020-07-08 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Obesity; Technology; Videoconferencing; mHealth; Behavior, Health
MeSH Terms: conditions — Obesity; Health Behavior | interventions — Telemedicine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Amulet only: As per usual care participants will receive an eHealth (Amulet + videoconferencing) intervention over a 16 week period of time.
  Interventions: Behavioral: eHealth
- Amulet/Fitbit: As per usual care participants will receive an eHealth (Amulet/Fitbit + videoconferencing) intervention over a 16 week period of time.
  Interventions: Behavioral: eHealth
- Fitbit only: As per usual care participants will receive an eHealth (Fitbit + videoconferencing) intervention over a 16 week period of time.
  Interventions: Behavioral: eHealth

INTERVENTIONS:
Behavioral: eHealth — Intervention Description: The pilot comprises of five components listed below which provide access to specialty obesity care to rural obese adults, and enhance it with technology (telehealth and remote monitoring): Team-based care; medical plan, nurses, psychologists, dietician, Health coaching, Weekly coaching sessions , Messaging and Remote Monitoring

SUMMARY:
The national epidemic of obesity is associated with considerable morbidity, disability and early mortality.

Conventional weight loss programs beyond a primary care setting have the potential to reduce weight, but are difficult to access for adults with obesity in rural areas due to lack of transportation and access to specialty care. Routine intensive behavioral therapy, while effective, is often not supplemented with adjuncts that could be helpful in engaging participants in behavioral change. The overarching goal of this SYNERGY pilot project is to overcome barriers rural adults face by using video-conferencing to deliver specialty obesity care that otherwise is inaccessible to most adults faced with this disease. It also intends to use emerging mobile health (mHealth) technology which has shown considerable promise in providing motivational feedback. This proposal highlights T3/T4 translation bridging technologists, allied health staff, and clinicians in the development and implementation of new therapeutic modalities. The study aims to evaluate a telehealth-based health coaching program that is embedded in the Dartmouth-Hitchcock Weight and Wellness Center that integrates novel remote monitoring technology in effecting behavioral change using Amulet, a Dartmouth Computer Science developed mHealth device over a 16-week period. First, the feasibility and accessibility of an eHealth-delivered health coaching obesity intervention using remote monitoring and video-conferencing (Aim 1) will be evaluated. The potential effectiveness of achieving the primary outcome of 5% weight loss, with secondary outcomes of improved physical function and self reported health (Aim 2) will be ascertained. The intervention's impact on implementation outcomes of workflow, adoption, and organizational change that could affect further scalability and generalizability in other high-risk population groups (Aim 3) will be assessed. These preliminary findings will be used in a future competitive application for an extramural R01 designed to assess the effectiveness of our intervention in achieving weight loss in rural obese adults. If successful, this application has the potential to redesign care using applied methods of telehealth translated to community-based, rural populations to facilitate behavioral change. The project also meets criteria of the NIH Strategic Plan for Obesity and the Institute of Medicine's need for Telehealth research.

ELIGIBILITY:
Inclusion Criteria:

* English speaking;
* Community-dwelling;
* Age 18-65 years;
* Obesity based on: BMI ≥30kg/m2 54;
* Participating in the DH-WWC health coach program;
* Access to home, high-speed internet with Wi-Fi;
* Medical clearance from their primary care provider;
* Provide voluntary, written consent;
* Require an EHR patient portal account and credentials ; -----If subjects do not have an account, one will be created for the purposes of this study

Exclusion Criteria:

* Unwilling to participate in the 16 week pilot or complete study measures;
* Individuals unwilling/unable to provide consent;
* A medical record diagnosis of dementia as intensive behavioral therapy and health coaching require the ability to complete questionnaires and change behavior, all of which may be challenging in individuals with cognitive impairment;
* Cognitive impairment measured by the 6-item Callahan screen, a brief and reliable six-item screening questionnaire with acceptable sensitivity (88.7%) and specificity (88.0%) in identifying individuals with cognitive impairment. Its diagnostic properties are comparable to the full Folstein Mini-Mental Status Examination in those scoring ≥3. This questionnaire can be administered by telephone or face-to-face interview and is being as an adjunct to medical record documentation of cognitive impairment;
* Life-threatening illness including those receiving palliative care or hospice services;
* Nursing facility or hospital admission in the past six months;
* Psychiatric diagnosis that would interfere with study participation and require significant modification to meet their needs such as major depressive disorder, substance abuse, suicidal ideation or severe mental illness (schizophrenia, bipolar disorder);
* History of bariatric surgery;
* American College of Sports Medicine contraindications to exercise57 including: a resting heart rate of >120bpm; Blood pressure >180/100mmHg; unstable angina;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will recruit 30 older motivated adults with obesity (aged 18-65 years). This study pilot will be based at the Dartmouth-Hitchcock (D-H) Weight and Wellness Center (DH-WWC) in Lebanon, NH. No randomization will be performed. Health coaches will deliver the intervention to participants
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2017-11-29 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2019-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John A Batsis, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Batsis JA, McClure AC, Weintraub AB, Sette D, Rotenberg S, Stevens CJ, Gilbert-Diamond D, Kotz DF, Bartels SJ, Cook SB, Rothstein RI. Barriers and facilitators in implementing a pilot, pragmatic, telemedicine-delivered healthy lifestyle program for obesity management in a rural, academic obesity clinic. Implement Sci Commun. 2020 Sep 30;1:83. doi: 10.1186/s43058-020-00075-9. eCollection 2020. PMID 33015640

RESULTS

PARTICIPANT FLOW:
Groups:
- Combined Group (Amulet/Fitbit): Combined group (Amulet/Fitbit) - Groups were combined because there was not enough data to analyze them separately
- Fitbit Only: Fitbit only as a remote monitoring device (in lieu of Amulet)
- Amulet Only: Amulet only device for remote monitoring
Period: Overall Study
Arm/Group | Combined Group (Amulet/Fitbit) | Fitbit Only | Amulet Only
Started | 8 | 20 | 9
Completed | 6 | 14 | 7
Not Completed | 2 | 6 | 2

BASELINE CHARACTERISTICS:
Groups:
- Combined Amulet/Fitbit: As per usual care participants will receive an eHealth (Amulet/Fitbit + videoconferencing) intervention over a 16 week period of time.
  eHealth: Intervention Description: The pilot comprises of five components listed below which provide access to specialty obesity care to rural obese adults, and enhance it with technology (telehealth and remote monitoring): Team-based care; medical plan, nurses, psychologists, dietician, Health coaching, Weekly coaching sessions , Messaging and Remote Monitoring
- Total: Total of all reporting groups
Arm/Group | Combined Amulet/Fitbit | Amulet Only | Fitbit Only | Total
Number analyzed (Participants) | 8 | 9 | 20 | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 9 | 20 | 37
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.4 (12.5) | 49.4 (10.3) | 45.1 (12.1) | 46.9 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16 | 32
  Male | 0 | 1 | 4 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 8 | 9 | 20 | 37
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 9 | 20 | 37

OUTCOME MEASURES:

1. Primary Outcome: Completion Rate: Number of Participants Completing the Intervention
Description: Completion/ Feasibility: The following rates will be computed: screened for inclusion; eligibility; enrollment; completion; assessment. We will assess entry criteria (reasons for dropout/non-adherence) and time to collect data. Enrollment success will be defined as 30 patients. Adequate retention is defined as a dropout rate of <20%. Completion of >80% of post-study measures will be defined as adequate. Attending >80% of sessions will be considered acceptable. Staff will track equipment, software or technical issues (malfunctions, data loss, hardware) in a journal.
Time Frame: 16 weeks
Population: Total completers
Measure: Count of Participants; unit: Participants
Groups:
- Combined Amulet/Fitbit: As per usual care participants will receive an eHealth (Amulet + videoconferencing) intervention over a 16 week period of time.
  eHealth: Intervention Description: The pilot comprises of five components listed below which provide access to specialty obesity care to rural obese adults, and enhance it with technology (telehealth and remote monitoring): Team-based care; medical plan, nurses, psychologists, dietician, Health coaching, Weekly coaching sessions , Messaging and Remote Monitoring
- Fitbit Only: videoconferencing + fitbit
- Amulet Only: videoconferencing + amulet as a remote monitoring device
Arm/Group | Combined Amulet/Fitbit | Fitbit Only | Amulet Only
Number analyzed (Participants) | 6 | 14 | 7
Participants | 6 | 14 | 7

2. Primary Outcome: Acceptability
Description: Acceptability: Qualitative interviews will ensure the appropriateness of the pilot and its strengths/weaknesses. Participants will answer questions on a scale from 0-5, where 5 = high acceptability of the program.
Time Frame: 16 Weeks
Population: On a scale of 0 (very disatisfied) to 5 (very satisfied) regarding the acceptability of the intervention
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Combined Amulet/Fitbit | Amulet Only | Fitbit Only
Number analyzed (Participants) | 6 | 7 | 14
score on a scale | 4 [4 to 5] | 4 [3 to 5] | 5 [4 to 5]

3. Secondary Outcome: Change in Weight
Description: Weight will be measured using a Seca 770 analyzer (in clinic) and by the Omron HBF-514 (at home remotely). Weight Loss (change in weight)
Time Frame: Baseline/16 weeks
Measure: Mean (Standard Deviation); unit: weight change (kg)
Groups:
- Amulet: As per usual care participants will receive an eHealth (Amulet + videoconferencing) intervention over a 16 week period of time.
  eHealth: Intervention Description: The pilot comprises of five components listed below which provide access to specialty obesity care to rural obese adults, and enhance it with technology (telehealth and remote monitoring): Team-based care; medical plan, nurses, psychologists, dietician, Health coaching, Weekly coaching sessions , Messaging and Remote Monitoring
Arm/Group | Combined Amulet/Fitbit | Fitbit Only | Amulet
Number analyzed (Participants) | 6 | 14 | 7
weight change (kg) | -0.47 (2.77) | -3.06 (3.63) | -2.51 (2.16)

4. Secondary Outcome: Change in 6 Minute Walk
Description: 6-Minute Walk (6MWT) is a cardiovascular fitness surrogate measuring distance (normal 400-700m) related to function. A clinically important difference or change is 50-55m
Time Frame: Baseline/16 weeks - pre/post change - increase = longer distance
Population: 2 participants in combined amulet/fitbit group were unable to perform assessment
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Combined Amulet/Fitbit | Amulet Only | Fitbit Only
Number analyzed (Participants) | 4 | 7 | 14
meters | 111.25 (27.8) | 227.14 (140.14) | -45.67 (180.5)

5. Secondary Outcome: Diet Change
Description: The Rapid Eating Assessment for Participants (REAPS) is a 16 item survey (score 13-39) of diet habits. Higher scores = higher diet quality. Positive score = better diet quality
Time Frame: Baseline/16 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Combined Amulet/Fitbit | Fitbit Only | Amulet
Number analyzed (Participants) | 6 | 14 | 7
units on a scale | 3.17 (4.71) | 2.42 (4.11) | 2.85 (2.91)

6. Secondary Outcome: Subjective Health
Description: The 10-question, non-proprietary Patient Reported Outcomes Measurement Information Systems General Health-10 (PROMIS) captures physical, mental and social aspects of quality of life. Positive change scores = improved health. The score ranges from 0-100, 50 is the population mean, 10 consists of 1SD, and higher scores equate better health.
Time Frame: Baseline/16 weeks - Change
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Combined Amulet/Fitbit | Fitbit Only | Amulet
Number analyzed (Participants) | 6 | 14 | 7
units on a scale | 2.58 (6.11) | 4.54 (4.38) | 5.6 (6.8)

7. Secondary Outcome: Readiness to Change
Description: The University of Rhode Island Change Assessment is a 12 item questionnaire assessing one's stages of change based on contemplation, action, maintenance and pre-contemplation.. The range of scores from -2 to +14. Higher scores indicate higher readiness to change
Time Frame: 16 weeks
Population: higher score indicates higher readiness to change. The range of scores from -2 to +14. Higher scores indicate higher readiness to change
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Amulet/Fitbit | Fitbit Only | Amulet
Number analyzed (Participants) | 6 | 14 | 7
score on a scale | 10.22 (1.31) | 9.64 (2.33) | 10.3 (1.9)

8. Secondary Outcome: Willingness to Pay
Description: Patient Perception of Value: Two questions will assess Willingness to Pay (WTP) - whether they would pay for telemedicine delivery of the intervention in lieu of in-person travel time or cost.
Time Frame: 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Amulet/Fitbit | Amulet Only | Fitbit Only
Number analyzed (Participants) | 6 | 7 | 14
Participants
  Time: >60min | 0 | 1 | 3
  Time: <60min | 6 | 6 | 11
  Cost <$30: >60min | 5 | 7 | 11
  Cost <$30: <60min | 1 | 0 | 3

9. Other Pre Specified Outcome: Staff Adoption
Description: Staff Adoption: Haug's 12-item Measure of Evidence-Based Practice Adoption assesses stage of change, experience, attitudes, organization barriers and strategies to support evidence-based practices (1-5 point scale - strongly disagree to agree).
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Staff Adoption: quantitative scale of staff adoption - 12 questions, each ranging 1-5
Arm/Group | Staff Adoption
Number analyzed (Participants) | 8
units on a scale | 2.64 (0.49)

ADVERSE EVENTS:
Time Frame: study itself - 16weeks;
Description: All subjects were asked about potential adverse events by the study interventionists at each study visit
Arm/Group | Combined Amulet/Fitbit | Amulet Only | Fitbit Only
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/9 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/9 | 0/20
Other Adverse Events (participants affected / at risk) | 0/8 | 0/9 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-06): https://cdn.clinicaltrials.gov/large-docs/87/NCT03309787/Prot_SAP_000.pdf